CLINICAL TRIAL: NCT04301128
Title: Research Asistant in Deparment of Nursing
Brief Title: The Effect of Mobile Application on Subcutaneous Anti-TNF Drug Administration:Ankylosing Spondylitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Fusun Uzgor, Research Assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 80558721/261; AZ142 (Other: Eskisehir Osmnagazi University)
Record Dates: First submitted 2020-02-27; First posted 2020-03-10 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2020-09

CONDITIONS: Ankylosing Spondylitis; Spondylitis, Ankylosing
Keywords: anti-TNF; mobile application; nursing; ankylosing Spondylitis; drug administration
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): Patients in the experimental group were able to install and set up mobile application on android phones via Bluetooth and were informed about the sick android application. Patients were reminded and guided by subcutaneous anti-TNF drug treatments from mobile application. Both groups of patients were then assessed using face-to-face interviews for 6 months, 6 weeks after using the Subcutaneous Anti-TNF Treatment Questionnaire , BASDAI, ASQoL, BASFI scales.
  Interventions: Other: Experimental
- BOOKLET GROUP (Active Comparator): An anti-TNF drug administration training booklet were given to patients in the control group and were required to take advantage of the booklet on subcutaneous anti-TNF drug production. Both groups of patients were then assessed using face-to-face interviews for 6 months, 6 weeks after using the Subcutaneous Anti-TNF Treatment Questionnaire , BASDAI, ASQoL, BASFI scales. At the end of the study (twenty forth week) was applied to all patients.
  Interventions: Other: control

INTERVENTIONS:
Other: Experimental — Patients in the experimental group were educated and followed with an android based mobile application which contains the informations related to the disease, treatment and its complications, monitoring and cure and provides side effect tracking.
  Arms: EXPERIMENTAL GROUP
Other: control — Patients in the control group were informed same informations verbally and given an education book.
  Arms: BOOKLET GROUP

SUMMARY:
This study was carried out to develop an android mobile application for the subcutaneous (SC) anti-TNF drug administration of ankylosing spondylitis patients and to evaluate its effect on drug administration.

The universe of this experimental designed posttest control group research is consisted of patients prescribed subcutaneous anti-TNF drug due to ankylosing spondylitis in Eskişehir Osmangazi University Health, Application and Research Hospital Rheumatology Polyclinic between 15 December 2017 - 30 December 2019. The patients who constituted the sample of the study were assigned by lot to mobile application and the education booklet groups. The mobile application that includes follow-up and information related to disease information, anti-TNF drug application and management was transferred to mobile phones of patients in mobile application group via bluetooth technology and installed. The patients in the education booklet group were given an education booklet on disease information, antiTNF drug administration and management. In the study, patients were evaluated once before anti-TNF drug treatment and every 6 weeks during 6 months (4 times) after treatment. The data of the study were collected by means of an individual identification form, BASDAI, BASFI, ASQoL and Subcutaneous Anti-TNF Treatment Questionnaire .

DETAILED DESCRIPTION:
Ankylosing spondylitis is a chronic, inflammatory disease that affects the axial spine, causing progressive limitation on the spine and leading to a decrease in quality of life. Anti TNF drugs are frequently used in the treatment of ankylosing spondylitis and teaching activities in improving patient compliance and patient compliance are very important in the success of this treatment. This study was carried out to develop an android mobile application for the subcutaneous (SC) anti-TNF drug administration of ankylosing spondylitis patients and to evaluate its effect on drug administration.

The universe of this experimental designed posttest control group research is consisted of patients prescribed subcutaneous anti-TNF drug due to ankylosing spondylitis in Eskişehir Osmangazi University Health, Application and Research Hospital Rheumatology Polyclinic between 15 December 2017 - 30 December 2019. The patients who constituted the sample of the study were assigned by lot to mobile application and the education booklet groups. The mobile application that includes follow-up and information related to disease information, anti-TNF drug application and management was transferred to mobile phones of patients in mobile application group via bluetooth technology and installed. The patients in the education booklet group were given an education booklet on disease information, antiTNF drug administration and management. In the study, patients were evaluated once before anti-TNF drug treatment and every 6 weeks during 6 months (4 times) after treatment. The data of the study were collected by means of an individual identification form, BASDAI, BASFI, ASQoL and Subcutaneous Anti-TNF Treatment Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* are diagnosed with ankylosing spondylitis according to the New York modification criterias
* administer anti-TNF agent for the first or second time
* are 18 years old and had literacy
* have an android phone,
* can use the andriod phone,
* agree to participate in the work

Exclusion Criteria:

* refuse to participate in the study
* be young than 18 years old
* administer anti-TNF agent more than twice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
subcutaneous anti TNF-α drug administration was assesed by "Subcutaneous Anti-TNF Treatment Questionnaire " | 4 times in 6 months
  In this questionnaire, It is expected from patients to answer "no" or "I always administered it myself" to these questions: "How often was your medication administered by someone else?", "In the last 6 weeks, did you ever miss or forget your dose of medication?" and "Did you ever skip implementing your medication dose thinking that your illness is under control?" Furthermore, the mean scores of "Overall difficulty level in continuing SC anti-TNF drug treatment" and "Satisfaction level with anti-TNF drug treatment in the last 6 weeks" are expected to be high.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Özkaraman, Study Director — Eskisehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University Faculty of Health Sciences, Eskişehir, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided